CLINICAL TRIAL: NCT02514824
Title: MLN0128 in Recurrent/Metastatic Merkel Cell Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Robert I. Haddad, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-223
Record Dates: First submitted 2015-07-28; First posted 2015-08-04 (Estimated); Results first posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Merkel Cell Carcinoma
Keywords: recurrent merkel cell carcinoma; metastatic merkel cell carcinoma
MeSH Terms: conditions — Carcinoma, Merkel Cell | interventions — sapanisertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dose Level 1: MLN01283 3 mg (Phase 1) (Experimental): Phase 1 dose level 1 participants receive MLN01283 3 mg orally once daily of a 28 day cycle.
  Participants are treated indefinitely until disease progression, unacceptable toxicity or withdrawal for other reasons.
  Interventions: Drug: MLN0128
- Dose Level 2: MLN01283 4 mg (Phase 1) (Experimental): Phase 1 dose level 2 participants receive MLN01283 4 mg orally once daily of a 28 day cycle.
  Participants are treated indefinitely until disease progression, unacceptable toxicity or withdrawal for other reasons.
  Interventions: Drug: MLN0128
- Dose Level 3: MLN01283 5 mg (Phase 1) (Experimental): Phase 1 dose level 3 participants receive MLN01283 5 mg orally once daily of a 28 day cycle.
  Participants are treated indefinitely until disease progression, unacceptable toxicity or withdrawal for other reasons.
  Interventions: Drug: MLN0128
- MLN01283 RP2D (Phase 2) (Experimental): Phase 2 participants receive MLN01283 at the recommended phase 2 dose (RP2D) orally once daily of a 28 day cycle.
  Participants are treated indefinitely until disease progression, unacceptable toxicity or withdrawal for other reasons.
  Interventions: Drug: MLN0128

INTERVENTIONS:
Drug: MLN0128 — Investigational mTOR kinase inhibitor
  Other Names: INK128

SUMMARY:
This research study is studying a targeted therapy as a possible treatment for merkel cell carcinoma.

- The name of the study intervention involved in this study is: MLN0128.

DETAILED DESCRIPTION:
This is a phase I/II clinical trial. A phase I clinical trial tests the safety of an investigational intervention and also tries to define the appropriate dose of the investigational intervention to use for further studies. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved MLN0128 as a treatment for any disease.

MLN0128 may prevent tumor cells from dividing and growing by selectively and potently inhibiting a chemical, mTOR kinase, which regulates cell growth and survival.

Patients with merkel cell carcinoma have been observed to sometimes carry genetic alterations in their tumor cells which may make the cancer more sensitive to inhibition by MLN0128. In this research study,the investigators are studying the usefulness of MLN0128 in merkel cell carcinoma cases.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic or recurrent MCC confirmed by histology
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as > 10 mm with spiral CT scan (see section 10 for the evaluation of measureable disease). Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented
* Age 18 years or older
* ECOG performance status ≤ 2
* Participants must have normal organ and marrow function
* Female patients who:

  * Are postmenopausal for at least 1 year before the screening visit

    --- OR
  * Are surgically sterile --- OR
* If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time
* Male patients, even if surgically sterilized (ie, status post-vasectomy), who:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, or
  * Agree to completely abstain from heterosexual intercourse
  * Treatment with strong CYP2C19, CYP3A4, and CYP2C9 inhibitors and/or inducers
  * Tissue for correlative studies must be available (paraffinized or frozen)
  * Ability to swallow oral medications and maintain an empty stomach state for 2 hours prior to the MLN0128 dose and for 1 hour following administration
  * Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Participants who have had chemotherapy or radiotherapy within 2 weeks prior to entering the study
* The subject has active brain metastases or epidural disease
* Participants who are receiving any other investigational agents within 14 days before the first dose of study drug
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations
* Female patients who are both lactating and breastfeeding or have a positive serum pregnancy test during the screening period or a positive urine pregnancy test on Day 1 before first dose of study drug
* Manifestations of malabsorption due to prior gastrointestinal (GI) surgery, GI disease, or for an unknown reason that may alter the absorption of MLN0128
* Poorly controlled diabetes mellitus
* History of any of the following within the last 6 months prior to study entry:

  * Ischemic myocardial event
  * Ischemic cerebrovascular event
  * Requirement for inotropic support (excluding digoxin) or serious (uncontrolled) cardiac arrhythmia
  * Placement of a pacemaker for control of rhythm
  * New York Heart Association (NYHA) Class III or IV heart failure
  * Pulmonary embolism
* Significant active cardiovascular or pulmonary disease at the time of study entry, including:

  * Uncontrolled high blood pressure
  * Pulmonary hypertension
  * Uncontrolled asthma
  * Significant valvular disease; severe regurgitation or stenosis
  * Medically significant (symptomatic) bradycardia
  * History of arrhythmia requiring an implantable cardiac defibrillator
  * Baseline prolongation of the rate-corrected QT interval (QTc)
* Initiation of treatment with hematopoietic growth factors, transfusions of blood and blood products, or systemic corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Haddad, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. Cumulative data will be posted here and published.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled from October 2015 through March 2017.
Groups:
- Dose Level 1: MLN01283 3 mg (Phase 1): Phase 1 dose level 1 participants receive MLN01283 3mg orally once daily of a 28 day cycle.
  Participants are treated indefinitely until disease progression, unacceptable toxicity or withdrawal for other reasons.
Period: Overall Study
Arm/Group | Dose Level 1: MLN01283 3 mg (Phase 1) | Dose Level 2: MLN01283 4 mg (Phase 1) | Dose Level 3: MLN01283 5 mg (Phase 1) | MLN01283 RP2D (Phase 2)
Started | 4 | 5 | 0 | 0
Evaluable for Dose-limiting Toxicity | 3 | 5 | 0 | 0
Completed | 3 | 4 | 0 | 0
Not Completed | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Dose-Limiting Toxicity | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population is comprised of all enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1: MLN01283 3 mg (Phase 1) | Dose Level 2: MLN01283 4 mg (Phase 1) | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Continuous [Median (Full Range); unit: years] | 69 [52 to 74] | 69 [60 to 75] | 69 [52 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 5 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: MLN01283 Maximum Tolerated Dose (MTD) [Phase I]
Description: The MLN01283 MTD is determined by the number of participants who experience a dose limiting toxicity (DLT). See subsequent primary outcome measure for the DLT definition. The MTD is defined as the highest dose at which fewer than one-third of patients experience a DLT. If no DLTs are observed, the MTD is not reached but the highest dose received may be the Recommended Phase II Dose (RP2D).
Time Frame: The observation period for DLT evaluation was the first 28 days (cycle 1) of treatment.
Population: All P1 participants who received at least one dose of the study drug were evaluable for the DLT analysis. Participants who discontinued study treatment prior to end of cycle 1 for reason other than dose-limiting toxicity were replaced.
Measure: Number; unit: mg
Groups:
- All Phase 1 Participants: Phase 1 participants received MLN01283 according to the established dose escalation schedule.
  Participants are treated indefinitely until disease progression, unacceptable toxicity or withdrawal for other reasons.
Arm/Group | All Phase 1 Participants
Number analyzed (Participants) | 8
mg | 3

2. Primary Outcome: Dose Limiting Toxicity (DLT) [Phase I]
Description: A DLT was defined as an adverse event (AE) assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications meets any of the following criteria including but not limited to: grade (G) 4-5 AEs, G3 thrombocytopenia, neutropenia, AST, ALT, serum creatinine or total bilirubin 2 to 3 x upper limit normal (ULN), aymptomatic amylase and/or lipase lasting >7 consecutive days; febrile neutropenia; G3 cardiac, hyperglycemia, mood alteration; G2 pancreatitis; G2 hyperglycemia unresolved within 14 days; G2 mood alteration unresolved in 14 days despite medical treatment; Dose interruption >21 days due to G2 dematologic; one grade level increase neurotoxicity.
Time Frame: The observation period for DLT evaluation was the first 28 days (cycle 1) of treatment.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: MLN01283 3 mg (Phase 1) | Dose Level 2: MLN01283 4 mg (Phase 1)
Number analyzed (Participants) | 3 | 5
Participants | 0 | 2

3. Post Hoc Outcome: Number of Participants With Objective Response (OR) [Phase 1]
Description: Objective response is defined as achieving complete response (CR) or partial response (PR) on treatment based on RECIST 1.1 criteria. For target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD.
Time Frame: Assessed on treatment and for this study cohort the longest treatment duration was approximately 4 months in each dose level 1 and 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: MLN01283 3 mg (Phase 1) | Dose Level 2: MLN01283 4 mg (Phase 1)
Number analyzed (Participants) | 4 | 5
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Assessed on treatment and for this study cohort the longest treatment duration was approximately 4 months in each dose level 1 and 2.
Description: Serious AEs (SAE) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher. All remaining AEs are classified as Other AEs (OAE) including grade 3 or higher events with treatment-attribution of unlikely and unrelated plus all grade 1 and 2 events. Maximum grade toxicity by type was then calculated within SAE and OAE datasets. No further data is available to specify classification of other beyond the general term.
Arm/Group | Dose Level 1: MLN01283 3 mg (Phase 1) | Dose Level 2: MLN01283 4 mg (Phase 1)
All-Cause Mortality (participants affected / at risk) | 3/4 | 3/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 3/5
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1: MLN01283 3 mg (Phase 1) (N=4) | Dose Level 2: MLN01283 4 mg (Phase 1) (N=5)
Nausea (Gastrointestinal disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1: MLN01283 3 mg (Phase 1) (N=4) | Dose Level 2: MLN01283 4 mg (Phase 1) (N=5)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 2
Bladder spasm (Renal and urinary disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
CPK increased (Investigations) | 0 | 1
Creatinine increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 2
Dizziness (Nervous system disorders) | 0 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Fall (General disorders) | 0 | 1
Fatigue (General disorders) | 3 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Headache (Nervous system disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 2
Hyponatremia (Metabolism and nutrition disorders) | 1 | 2
Hypotension (Vascular disorders) | 0 | 2
Infections and infestations - Other (Infections and infestations) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 4
Pain (General disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Upper respiratory infection (Infections and infestations) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Urinary urgency (Infections and infestations) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2
Weight loss (Investigations) | 1 | 3

LIMITATIONS AND CAVEATS:
The study did not proceed to phase 2 due to slow accrual and lack of efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2016-03-18): https://cdn.clinicaltrials.gov/large-docs/24/NCT02514824/Prot_000.pdf